CLINICAL TRIAL: NCT00512486
Title: A Multi-Center, Open-Label, Single Administration, Sequential Dose Escalation of BIW-8405/MEDI-563 in Subjects With Mild Asthma
Brief Title: A Sequential Dose-Escalation Study in Subjects With Mild Asthma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Responsible Party: Lenny Smith, Senior Clinical Progam Manager, MedImmune Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: MI-CP158
Record Dates: First submitted 2007-08-06; First posted 2007-08-07 (Estimated); Last update posted 2008-11-27 (Estimated); Status verified 2008-11

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — benralizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Active Comparator): MEDI-563
  Interventions: Biological: MEDI-563

INTERVENTIONS:
Biological: MEDI-563 — BIW-8405/MEDI-563 administered at one of five dose levels:
  * 0.03 mg/kg intravenous injection
  * 0.1 mg/kg intravenous injection
  * 0.3 mg/kg intravenous injection
  * 1.0 mg/kg intravenous injection
  * 3.0 mg/kg intravenous injection
  Following the -3.0 mg/kg dose level,
  BIW-8405/MEDI-563 administered at one of two lower dose levels:
  0.003 mg/kg intravenous injection 0.0003 mg/kg intravenous injection

SUMMARY:
The primary objective of this study is to investigate the safety of administration of this drug by increasing doses to male and female adult subjects with mild asthma.

DETAILED DESCRIPTION:
The primary objective of this study is to investigate the safety of administration of BIW-8405/MEDI-563 in increasing doses to male and female adult subjects with mild asthma.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged 18 through 45 years in good general health other than asthma that is consistent with the definition of mild (intermittent or persistent) asthma by the 2002 Expert Panel report of the NAEPP: Night time symptoms no more than once weekly and day time symptoms <1 per day; lung function, FEV1 or PEF ≥ 80% of predicted value and PEF variability ≤ 30%. Note: the Principal Investigator must determine that the subject's asthma is consistent with this definition e.g., it is not required for the Investigator to obtain historical PEF values to calculate variability.
2. Subjects with a PC20 methacholine of ≤ 8 mg/mL at Visit 1 (required for subjects in Cohorts 5-7) or documented within 6 months prior to Visit 1 (for subjects in Cohorts 1-4).3. Subjects who have provided written informed consent. Written informed consent must be obtained prior to performing any study related procedures.

4. Subjects who are considered by the Principal Investigator to be otherwise healthy, as judged by the absence of clinically significant diseases or clinically significant abnormal laboratory values that would confound interpretation of the study.

5. Women must be post menopausal, surgically sterile or willing to use birth control for the duration of the study. Birth control may include double barrier methods (e.g., condom with spermicide, hormonal contraceptives (provided they have been used regularly for at least 3 menstrual cycles) or IUD (provided it has remained in situ for at least three menstrual cycles).

Exclusion Criteria:

1. All asthmatic subjects who have received topical steroids (except nonprescription topical steroids for dermatologic conditions) within 6 months prior to Visit 1 will be excluded.
2. Any subject requiring a prescription medication, other than contraceptives or a β2 agonist (eg, albuterol) or anticholinergic agent (eg, ipratropium) for the treatment of mild asthma during the study. Subjects taking nonprescription medications must be willing and able to refrain from their use during the inpatient period of the study.
3. Any subject who has smoked cigarettes or cigars within one year prior to Visit 2 or has smoked for > 5 pack/years.
4. Any subject with documented evidence of Hepatitis B virus, HIV or hepatitis C virus (HCV) infection.
5. Any subject who has been documented as being Mantoux (PPD) positive.
6. Any subject having a parasitic infection at any time in the past or intending to travel to an area where parasitic infections are endemic.
7. Any subject with any condition resulting in an increased eosinophil count (except asthma) at screening.
8. Any subject with a Body Mass Index less than 15 kg/m2 or greater than 30 kg/m2 at Visit 1.
9. Any subject with a documented history of disorders of the immune system (except asthma) at any time.
10. Any subject with a clinically relevant abnormality of any laboratory parameter during the screening period (except eosinophilia due to asthma).
11. Any subject who has participated in any other study of an investigational product within either 30 days or 10 half lives (if known) prior to Visit 2, whichever is longer.
12. Any subject with a history of dependence on alcohol or drugs of abuse or with a positive drug screen at Visit 1.
13. Any subject with known sensitivity to any constituent of BIW-8405/MEDI-563 or any other IL-5 receptor antagonist.
14. Any subject with a history of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, or neurological disorder that is capable of altering the metabolism or elimination of drugs or that constitutes a risk factor when taking the study medication.
15. Any subject with a clinically significant relevant deviation from normal in physical examination, electrocardiography, or clinical laboratory tests, as determined by the Principal Investigator.
16. Any subject who has donated blood or in any other way had a loss of blood volume greater than 450 mL within 30 days before beginning the study injection.
17. Any subject who is unwilling to reside in the clinic during the study period or is unwilling to cooperate fully with the Principal Investigator or designee.
18. Pregnant females will be excluded from study participation.
19. Any subject who plans to undergo elective surgery within 4 weeks before Visit 2 (Day 0) through the end of the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2006-11; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the overall incidence of adverse events reported in each dose group. | Day 84

SECONDARY OUTCOMES:
Laboratory assessments of safety (hematology, biochemistry and urinalysis), assessments of immunogenicity, vital signs, physical examinations, and ECGs. | Day 84
Safety will also be assessed by measurement of T-cell, B-cell, and NK counts using fluorescence activated cell sorter (FACS) technology. | Day 84
Secondary pharmacological endpoints will include assessments of eosinophil counts in peripheral blood, FENO, and ECP. | Day 84

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Molfino, M.D., Study Director — MedImmune LLC
Locations (3):
- United States (3):
  - Jewish Medical and Research Center, Denver, Colorado
  - Northeast Medical Research Associates, Inc., North Darthmouth, Massachusetts
  - Allergy-Asthma-K4, Madison, Wisconsin